CLINICAL TRIAL: NCT01791270
Title: Expression of Maxi-k+ Channel β1 Subunit in Peripheral Leukocytes, Blood Pressure Values and the Presence of Endothelial Dysfunction in Patients With Obstructive Sleep Apnea
Brief Title: Obstructive Sleep Apnea (OSA), Hypertension , β1 Subunit of Maxi-k+ Channel and Cardiovascular Risk
Acronym: OSAS
Status: Completed | Type: Observational
Sponsor: Angeles Sanchez Armengol (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Sponsor-Investigator, Angeles Sanchez Armengol, MD PhD, Sociedad Española de Neumología y Cirugía Torácica
Organization: Sociedad Española de Neumología y Cirugía Torácica (Other)
Other Study IDs: P09-CTS-4971
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Hypertension; β1 Subunit of Maxi-k+Channel; Cardiovascular Risk
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — Continuous Positive Airway Pressure; Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Periferical blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSA versus Control subjects.: sleep apnea-hypopnea syndrome and control
- OSA patients before and after treatment, CPAP: Continuous positive pressure CPAP
  Interventions: Device: Continuous positive airway pressure (CPAP) therapy

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) therapy — Device: CPAP accordingly to the normal therapy in daily practice. In the group of 61 patients with OSA: we compared the results before and after three months of correct treatment with CPAP.
  First, an automatic continuous positive airway pressure device (autoCPAP REMstar) was used to evaluate the pressure titration by night registration at patient home. AutoCPAP gets complete information about the optimum level to be set as therapeutic (CPAP pressure).
  The patient has been reevaluated periodically in the outpatient Sleep Unit to verify proper adaptation and compliance of CPAP.
  We considered a proper compliance when patients used CPAP ≥ 4 hours/day. This data has been extracted from the counter included in the CPAP compressor.
  Procedures:
  1. - Respiratory Polygraphy
  2. - Ambulatory Blood Pressure Monitoring
  3. - Endothelial dysfunction, by determining the hyperaemic response to ischemia using a Laser-Doppler flowmeter.
  4. - ß1en subunit expression in peripheral blood leukocytes.
  Groups: OSA patients before and after treatment, CPAP

SUMMARY:
To describe the relationship between OSA and clinical Hypertension (performing ABPM), endothelial dysfunction (performing flowmetry), and its relation at the basic research (determining the β1 subunit in Peripheral Leukocytes in peripheral blood). This relation between OSA and HTA has been evaluated in basal conditions and after modifying the pathophysiological role of OSA applying treatment with positive continues pressure (CPAP) during 3 months.

DETAILED DESCRIPTION:
Background: Several epidemiological studies have demonstrated that untreated OSA with continuous positive airway pressure, is related to high rates of cardiovascular morbidity and mortality, being HTA the most important cardiovascular morbidity associated with OSA. This relationship has been studied at three levels: clinical, subclinical and the basic research or molecular level. Most patients with OSA diagnosis have developed clinical hypertension and, because of the high prevalence of nocturnal hypertension in OSA, it would be essential to monitor blood pressure during sleep, using this device ambulatory blood pressure monitoring (ABPM). Regard to endothelial dysfunction, which can exist before irreversible vascular changes have occurred in the arterial wall (subclinical level) has been reported that patients with OSA have lower blood flow (measured by arterial flowmetry) and after treatment with CPAP, there is an improvement in endothelial function. At basic research level, in previous studies it has been observed that hypoxia down regulates the expression of Maxi-K+ Channel B1-subunit in smooth muscle cell and also in peripheral leukocytes. This channel is involved in the regulation of arterial vasodilation, being β1 subunit responsible for the vascular tone regulation. Basic research studies have shown the relationship between hypertension and ß1 subunit, describing that the expression of that unit decreases in hypertensive animal models. In a pilot study in OSA patients was suggested that ß1 subunit channel Maxi-K + could play an important role in vascular dysregulation of these patients. It has been also described a correlation between ß1 subunit level in vascular smooth muscle cells and its level in leukocytes.

Objective: To describe the relationship between OSA and hypertension from a clinical point of view (by performing ABPM), its relationship with endothelial dysfunction (by performing a flowmetry) and basic research level (by the determination of β1 subunit of the maxi-K channel +). This relationship between hypertension and OSA has been assessed at baseline condition in a group of OSA patients and a control group without OSA, and after changing the pathophysiological role of OSA treating with continuous positive pressure airway (CPAP) in the group of OSA patients.

Patients: Prospective study in which:

1. - We compared 61 patients with sleep apnea-hypopnea syndrome and 19 control subjects without OSA.
2. - In the group of 61 patients with OSA: we compared the results before and after three months of correct treatment with CPAP.

Measurements:

1. - Respiratory Polygraphy
2. - Ambulatory Blood Pressure Monitoring
3. - Endothelial dysfunction, by determining the hyperaemic response to ischemia using a Laser-Doppler flowmeter.
4. - ß1en subunit expression in peripheral blood leukocytes.

These procedures are described below:

1. - Respiratory Polygraphy:

   -Nocturnal cardiorespiratory polygraphy was performed in the "sleep laboratory of Medical-Surgical Unit of Respiratory Diseases". It has used a respiratory polygraph "Sibelhome plus"(trade name).

   We measured the following variables:
   * Oronasal Flow.
   * Snore: using laryngotracheal microphone.
   * Thoracoabdominal-Effort: by two bands effort sensors placed at the level of the chest and abdomen.
   * Arterial oxygen saturation (SaO2): Flexible digital pulse oximeter.
   * Body-position sensor.

   The records are stored in a specific database and analysis was carried out manually. The events are defined
   * Apnea: absence of oronasal airflow for ≥ 10 sec.
   * Hypopnea: oronasal flow decrease ≥ 50% from baseline for ≥ 10 seconds, accompanied by desaturation.

   We calculated the following parameters:
   * AHI: total number of apnea + hypopnea / hour check. When AHI is <5 was considered negative for OSA and when AHI WAS ≥ 15, OSA diagnosis was made.
   * Desaturation index (DI): total number of desaturations / hour check.
   * Basal and minimum-Saturation: automatic analysis obtained oximetry throughout the entire record.
   * Percentage of recording time with SaO2 <90% (CT90): automatic analysis obtained oximetry throughout the entire record.
2. - Ambulatory Blood Pressure Monitoring: The dispositive measures blood pressure automatically every 20 minutes for 24 hours. The records were obtained on a weekday and when the patient worked in shifts, it was made when the patients didn´t work at night.

   We collected the following variables:
   * 24hours systolic and diastolic blood pressure.
   * Medium blood pressure at day and night.
   * Standard deviation day and night blood pressure.
   * Percentage of high measured for 24 hours, and during periods of activity and rest.
   * BP variability (standard deviation of the mean).
   * 24-hour mean heart rate.
   * Average heart rate daytime.
   * Night Average heart rate.
3. - Endothelial dysfunction, by determining the hyperaemic response to ischemia using a Laser-Doppler flowmeter: The subject lay on the bed, and kept quiet 15-20 minutes. A cuff blood pressure measurement (uninflated) was placed on the arm and laser-Doppler device in the forearm. During 15 minutes the system measured basal situation and after that the cuff rapidly swelled over 20mmHg of the systolic blood pressure during for 4 minutes. During this period the system monitor showed perfusion units and at the end of this period the cuff was suddenly deflated and the monitor revealed a rise above the pre-ischemia in perfusion units.

   The software performed two types of analysis:
   * General analysis: where reported the initial value, maximum value, percentage change from the first to last value or maximum slope of the curve or slope and area under the curve.
   * Adjusted Analysis: It was estimated biological zero, peak flow, hyperemia area, time to maximum hyperemia, time to reach the half-maximal hyperemia and latency.
4. - ß1 subunit expression in peripheral blood leukocytes: Performing the level of β1 subunit of Maxi-K + channel expression in peripheral blood leukocytes. Extraction total RNA from leukocytes following the instructions QIAamp RNA Blood Mini kit.

From these cells was performed the expression level of β1 subunit by quantitative RT-PCR technique. For reverse transcription of RNA using the Superscript III First-kit Starnd Synthesis System (trade name). For quantitative PCR we used the ABI PRISM equipment 7500 Sequence Detection System (Applied Biosystems), using the reagents Sybr Green PCR Master Mix or TaqMan probes, following the protocols indicated by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* The control group was defined as "absence of OSA"(apnea-hypopnea index (AHI) in cardiorespiratory polygraphy <5).
* The "OSA" group was defined as OSA symptoms + an AHI ≥ 15 in cardiorespiratory polygraphy

Exclusion criteria:

* Awaking hypoxemia (PO2 in arterial blood gas <70 mmHg) or arterial saturation <90% in digital pulse oximetry.
* Treated hypertensive patients who were not well controlled at the time of inclusion: change of HTA treatment in the previous 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group of OSA patients and a control group without OSA
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement in blood pressure parameters, in vascular endothelial function and in levels of β1 subunit expression of Maxi-K + channel in patients with OSA after treatment with CPAP | 3 months
  Primary Outcome Measure: Look at the difference in OSA and control subjects between the parameters that measure blood pressure in AMBP, the reactive hyperemia test for ischemia flowmetry technique and the expression levels of ß1 subunit of the Maxi-K + channel in peripheral blood leukocytes.
  In OSA group patients after three months of correct treatment with CPAP, the goal is to find:
  * Improvement in blood pressure parameters (ambulatory blood pressure).
  * Improved parameters expressing vascular endothelial function at subclinical level (recorded by laser-Doppler flowmetry).
  * Improvement in levels of β1 subunit expression of Maxi-K + channel in peripheral blood leukocytes (basic).

CONTACTS AND LOCATIONS:
Overall Officials: Angeles Sánchez Armengol, Md PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío

REFERENCES:
- [Derived] Caballero-Eraso C, Munoz-Hernandez R, Asensio Cruz MI, Moreno Luna R, Carmona Bernal C, Lopez-Campos JL, Stiefel P, Sanchez Armengol A. Relationship between the endothelial dysfunction and the expression of the beta1-subunit of BK channels in a non-hypertensive sleep apnea group. PLoS One. 2019 Jun 19;14(6):e0217138. doi: 10.1371/journal.pone.0217138. eCollection 2019. PMID 31216297